CLINICAL TRIAL: NCT05307432
Title: A Safety Planning Intervention and Follow-up Telehealth Service Model for Suicidal Individuals in Emergency Department Settings
Brief Title: Safety Planning Intervention Telehealth Service Model in Emergency Departments
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 850636; 1P50MH127511-01 (NIH)
Record Dates: First submitted 2022-03-02; First posted 2022-04-01 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Suicide; Suicidal Ideation
Keywords: Safety Planning; Emergency Department; Risk Assessment; Follow-up Contact; Implementation Strategies; Telehealth
MeSH Terms: conditions — Suicide; Suicidal Ideation; Emergencies

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster-randomized controlled design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (Active Comparator): ED staff deliver SPI+ (Safety Planning Intervention plus 2 or more post-discharge telephone calls) to suicidal patients who are not admitted to an inpatient unit.
  Interventions: Behavioral: SPI+ Delivered by ED Staff
- Suicide Prevention Consultation Center (Experimental): ED staff refer suicidal patients not admitted to an inpatient unit to the off-site Suicide Prevention Consultation Center (SPCC). SPCC clinicians will deliver SPI+ (Safety Planning Intervention plus 2 or more post-discharge telephone calls) to patients via telehealth.
  Interventions: Behavioral: SPI+ Delivered by SPCC Clinicians

INTERVENTIONS:
Behavioral: SPI+ Delivered by ED Staff — ED staff will deliver SPI+ (Safety Planning Intervention plus follow-up phone calls) to patients at risk for suicide in the ED who are not admitted to an inpatient unit.
  Arms: Enhanced Usual Care
Behavioral: SPI+ Delivered by SPCC Clinicians — The Suicide Prevention Consultation Center (SPCC) will be located external to the Emergency Department (ED). ED staff will be able to refer patients at risk for suicide to the SPCC. Licensed and credentialed mental health clinicians will deliver SPI+ (Safety Planning Intervention plus follow-up phone calls) via telehealth to patients at risk for suicide in the ED who are not admitted to an inpatient unit.
  Arms: Suicide Prevention Consultation Center

SUMMARY:
The purpose of this study is to evaluate the effectiveness and implementation of a suicide prevention strategy delivered via telehealth in Emergency Departments. We will compare implementation of the Safety Planning Intervention plus follow-up calls (SPI+) delivered by Emergency Department (ED) staff to SPI+ delivered via ED referral to an off-site Suicide Prevention Consultation Center (SPCC).

DETAILED DESCRIPTION:
Individuals at high risk for suicide often present to acute care settings, such as emergency departments (EDs), and then typically are hospitalized or referred for outpatient mental health treatment. Patients are at increased risk of suicide attempts and suicide following an ED visit and nearly half do not attend outpatient treatment. Brief, evidence-based clinical interventions, such as the Safety Planning Intervention with post-discharge telephone follow-up (SPI+), can reduce suicide risk, decrease hospitalizations, and increase engagement in outpatient services for suicidal patients discharged from the ED. Leveraging insights from implementation science and collaborative care, we propose a model in which ED staff will connect patients at risk for suicide to ED-credentialed mental health clinicians who are located external to the ED. These off-site clinicians will provide SPI+ via telehealth for ED patients prior to discharge and provide follow-up services after ED discharge as part of an innovative Suicide Prevention Consultation Center (SPCC). All participating EDs will begin in the Enhanced Usual Care phase, in which ED staff will deliver SPI+ to suicidal patients. EDs will then be randomized in pairs to begin referral to the SPCC in 3 month intervals. We will also conduct a cost evaluation to help determine scalability and sustainability.

ELIGIBILITY:
Aim 1/Aim 3:

Inclusion Criteria:

* ED visit at one of our participating sites for a suicide-related event or determined to be at risk for suicide per the Electronic Health Record (EHR) and ED clinical staff
* 18 years of age or older
* Not admitted to an inpatient hospital following the index ED visit as documented in the EHR

Exclusion Criteria:

- Inpatient admission following the index ED visit per the EHR

Aim 2:

Inclusion Criteria:

* ED clinician or leader at one of our participating sites, or ED patient who was referred to the SPCC
* 18 years of age or older
* Able to communicate in English
* Willing to give informed consent

Exclusion Criteria:

* Patients who are at imminent risk of suicide or acutely psychotic at the time of the interview, requiring emergency services and/or precluding ability to provide informed consent
* Patients without a phone for contact

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2814 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Suicide Behavior Composite | 6 months after index ED visit
  Number of patients who had a documented suicide attempt or death by suicide
Outpatient Treatment Engagement - Count | 6 months after index ED visit
  Number of behavioral healthcare visits following discharge from index ED visit
Outpatient Treatment Engagement - Type | 6 months after index ED visit
  Types of behavioral healthcare visits following discharge from index ED visit
Safety Planning Intervention Scoring Algorithm (SPISA) | At index ED visit
  Fidelity of written safety plans post-discharge from index ED visit
Fidelity of Follow-up Calls | 1 month after index ED visit
  Number of patients who had 2 or more follow-up calls post-discharge from index ED visit
Reach/Penetration of Safety Plans | At index ED visit
  Proportion of patients with a completed safety plan documented in the medical record out of all patients identified as at risk for suicide by the ED staff
Reach/Penetration of Follow-up Calls | 1 month after index ED visit
  Proportion of patients who receive 2 or more telephone follow-up attempts out of all patients who received a safety plan

SECONDARY OUTCOMES:
Suicide-related ED Visits and Psychiatric Hospitalizations | 6 months after index ED visit
  Number of ED visits and/or inpatient psychiatric admissions for suicidal ideation/behavior
Suicide Attempts | 6 months after index ED visit
  Number of patients who had a documented suicide attempt
Adoption | At index ED visit
  Proportion of clinicians with eligible patients who refer the patient to the SPCC
Utilization of Screening of Suicide Risk Among ED Patients | At index ED visit
  Proportion of ED patients who received the Columbia Suicide Severity Rating Scale or equivalent evidence-based measure of suicide risk during index ED visit
Index ED Visit Inpatient Admission Disposition | At index ED visit
  Proportion of patients admitted for inpatient hospitalization out of all patients identified as at risk for suicide
Feasibility of SPCC | 9-12 months after ED crosses over to SPCC condition
  Will be assessed through semi-structured qualitative interviews with a randomly selected sample of clinicians, leaders, and patients, as well as by using the Feasibility of Intervention Measure (FIM)
Acceptability of SPCC | 9-12 months after ED crosses over to SPCC condition
  Will be assessed through semi-structured qualitative interviews with a randomly selected sample of clinicians, leaders, and patients, as well as by using the Acceptability of Intervention Measure (AIM)
Cost to Emergency Department of SPCC | After ED crosses over to SPCC condition (2.25 - 3 year range, average of 2.625 years)
  We will assess average personnel and non-personnel costs to Emergency Department practices of delivering SPCC and EUC strategies, using Time-Driven Activity-Based Costing
Cost to Emergency Department of EUC | Before ED crosses over to SPC condition (1 - 1.75 year range, average of 1.375 years)
  We will assess average personnel and non-personnel costs to Emergency Department practices of delivering EUC strategies, using Time-Driven Activity-Based Costing

CONTACTS AND LOCATIONS:
Overall Officials: Gregory K Brown, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States